CLINICAL TRIAL: NCT02456896
Title: Effect of Oxcarbazepine on Serum Brain Derived Neurotrophic Factor (BDNF) in Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM-NF/Pharm/14/19
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Bipolar Disorder
Keywords: Oxcarbazepine; Brain Derived Neurotrophic Factor; Bipolar disorder; Neuroprotection
MeSH Terms: conditions — Bipolar Disorder | interventions — Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy control (No Intervention): Twenty five (25) age and sex matched healthy individuals will serve as the control group. Control subjects will be evaluated at baseline only.
- Oxcarbazepine (Experimental): Twenty five (25) patients of bipolar mania will be prescribed oxcarbazepine for 4 weeks.
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine — After baseline assessments, patients in test group will be prescribed Tab. Oxcarbazepine (600mg/daily in two divided dose for 1 week followed by 900mg/daily in two divided dose for next 3 weeks).
  Arms: Oxcarbazepine

SUMMARY:
The present study has been designed to evaluate the change in serum BDNF level with oxcarbazepine monotherapy in bipolar disorder and to explore the possibility of its neuroprotective effect.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a chronic psychiatric illness of partially unknown pathophysiology. BD likely involves, at a molecular and cellular level, dysfunctions of critical neurotrophic, cellular plasticity and resilience pathways and neuroprotective processes. Abnormalities of neurotrophins (NTs) and other trophic factors orchestrate important alterations which could be implicated in the etiology of BD. As consistently reported in post-mortem studies, these modifications are generally associated with the disruption of distinct subregions and functions of the brain, one of which is the deregulation of neurotrophins.

NTs are capable of signaling neurons, glial cells and other cellular systems to enable survival, differentiation and growth. BDNF is one of the most studied and abundant NTs in the brain, which plays an important role in a variety of neural processes during the development of both animals and humans. Initially, BDNF is important for neurogenesis, neuronal survival, and normal maturation of neural development pathways. In the adult, BDNF is not only important for synaptic plasticity and dendritic growth, but also for long-term memory consolidation. Several studies have proved that BDNF is significantly reduced in manic, hypomanic or depressive stages of BD, whereas euthymic patients exhibit BDNF levels similar to healthy controls.

Rafael T. de Sousa et al have observed a significant increase in serum BDNF levels after 28 days of lithium monotherapy in patients with BD and suggested neuroprotective role of lithium due to its direct regulatory effect on BDNF. Oxcarbazepine is a commonly used mood stabilizer which has demonstrated comparable efficacy to divalproate sodium and better tolerability profile but till date there is no study on its effect on BDNF. The aim of the present study is to evaluate the change in serum BDNF level with oxcarbazepine monotherapy in bipolar disorder and to explore the possibility of its neuroprotective effect.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the diagnosis of bipolar affective disorder (by ICD-10 DCR) current episode mania without psychotic symptoms
* Patients aged 18-45 years, of either sex.
* Patients with baseline score > 20 on the Young Mania Rating Scale (YMRS).
* Patients who had not taken any treatment for at least 4 weeks before inclusion.

Exclusion Criteria:

* Patients with bipolar disorder (by ICD-10 DCR) presenting during depressive/euthymic/mixed episode.
* Patients who are already under treatment for the presenting conditions.
* Rapid cycling in the past 12 months.
* Previous history of refractoriness to carbazepine or oxcarbazepine.
* Patients with comorbid substance abuse or history of organicity
* Pregnant and nursing women, patients with history of major medical or neurological illness.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DEBASISH HOTA, MD, DM, Study Director — AIIMS, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Odisha, India

REFERENCES:
- [Background] Frey BN, Andreazza AC, Houenou J, Jamain S, Goldstein BI, Frye MA, Leboyer M, Berk M, Malhi GS, Lopez-Jaramillo C, Taylor VH, Dodd S, Frangou S, Hall GB, Fernandes BS, Kauer-Sant'Anna M, Yatham LN, Kapczinski F, Young LT. Biomarkers in bipolar disorder: a positional paper from the International Society for Bipolar Disorders Biomarkers Task Force. Aust N Z J Psychiatry. 2013 Apr;47(4):321-32. doi: 10.1177/0004867413478217. Epub 2013 Feb 14. PMID 23411094
- [Background] Mufson EJ, Kroin JS, Sendera TJ, Sobreviela T. Distribution and retrograde transport of trophic factors in the central nervous system: functional implications for the treatment of neurodegenerative diseases. Prog Neurobiol. 1999 Feb;57(4):451-84. doi: 10.1016/s0301-0082(98)00059-8. PMID 10080385
- [Background] Huang EJ, Reichardt LF. Neurotrophins: roles in neuronal development and function. Annu Rev Neurosci. 2001;24:677-736. doi: 10.1146/annurev.neuro.24.1.677. PMID 11520916
- [Background] Kaplan DR, Miller FD. Neurotrophin signal transduction in the nervous system. Curr Opin Neurobiol. 2000 Jun;10(3):381-91. doi: 10.1016/s0959-4388(00)00092-1. PMID 10851172
- [Background] Post RM. Role of BDNF in bipolar and unipolar disorder: clinical and theoretical implications. J Psychiatr Res. 2007 Dec;41(12):979-90. doi: 10.1016/j.jpsychires.2006.09.009. Epub 2007 Jan 18. PMID 17239400
- [Background] Cunha AB, Frey BN, Andreazza AC, Goi JD, Rosa AR, Goncalves CA, Santin A, Kapczinski F. Serum brain-derived neurotrophic factor is decreased in bipolar disorder during depressive and manic episodes. Neurosci Lett. 2006 May 8;398(3):215-9. doi: 10.1016/j.neulet.2005.12.085. Epub 2006 Feb 9. PMID 16480819
- [Background] Fernandes BS, Gama CS, Cereser KM, Yatham LN, Fries GR, Colpo G, de Lucena D, Kunz M, Gomes FA, Kapczinski F. Brain-derived neurotrophic factor as a state-marker of mood episodes in bipolar disorders: a systematic review and meta-regression analysis. J Psychiatr Res. 2011 Aug;45(8):995-1004. doi: 10.1016/j.jpsychires.2011.03.002. Epub 2011 May 6. PMID 21550050
- [Background] de Sousa RT, van de Bilt MT, Diniz BS, Ladeira RB, Portela LV, Souza DO, Forlenza OV, Gattaz WF, Machado-Vieira R. Lithium increases plasma brain-derived neurotrophic factor in acute bipolar mania: a preliminary 4-week study. Neurosci Lett. 2011 Apr 20;494(1):54-6. doi: 10.1016/j.neulet.2011.02.054. Epub 2011 Mar 6. PMID 21362460
- [Background] Kakkar AK, Rehan HS, Unni KE, Gupta NK, Chopra D, Kataria D. Comparative efficacy and safety of oxcarbazepine versus divalproex sodium in the treatment of acute mania: a pilot study. Eur Psychiatry. 2009 Apr;24(3):178-82. doi: 10.1016/j.eurpsy.2008.12.014. Epub 2009 Mar 25. PMID 19324530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: June 2015 to December 2015 Psychiatry outpatient department
Pre-assignment Details: Out of 40 bipolar mania patients screened, 12 patients were excluded as they did not meet the inclusion criteria and another three patients declined to participate. For recruitment of healthy controls, 35 subjects were screened and after exclusion of 10 subjects, 25 were included in the study.
Groups:
- Healthy Control: Twenty five (25) age and sex matched healthy individuals served as the control group.
Period: Overall Study
Arm/Group | Healthy Control | Oxcarbazepine
Started | 25 | 25
Completed | 19 | 21
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Oxcarbazepine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.44 (9.53) | 34.16 (9.89) | 34.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 20 | 20 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  India | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Brain Derived Neurotrophic Factor (BDNF)
Description: Serum BDNF was estimated by ELISA using human BDNF ELISA kit from Boster Biological Technology Co. Ltd., Pleasanton, CA.
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Healthy Control | Oxcarbazepine
Number analyzed (Participants) | 19 | 21
pg/ml | 23.1 (92.7) | 90.7 (85.0)

2. Secondary Outcome: Correlation Between Young Mania Rating Scale (YMRS) and Serum Brain Derived Neurotrophic Factor (BDNF)
Description: The YMRS total score ranges from 0 to 60 where higher scores indicate more severe mania.
  Spearman's rank correlation coefficient (Spearman's ρ) was calculated for measuring correlation between YMRS score and serum BDNF.
Time Frame: At baseline
Population: At baseline
Measure: Number; unit: Spearman's ρ
Arm/Group | Healthy Control | Oxcarbazepine
Number analyzed (Participants) | 25 | 25
Spearman's ρ | -0.59 | -0.59

ADVERSE EVENTS:
Time Frame: 7 months
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Arm/Group | Healthy Control | Oxcarbazepine
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes